CLINICAL TRIAL: NCT03684850
Title: Effect of Unloader Knee Brace and Biomechanical Footwear Device on Symptoms and Physical Function in Knee Osteoarthritis Patients - a Randomized Controlled Trial
Brief Title: Knee Brace and Biomechanical Footwear in the Treatment of Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Finland Hospital District (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnro 11U/2015
Record Dates: First submitted 2017-01-30; First posted 2018-09-26 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2019-07

CONDITIONS: Osteoarthritis,Knee
Keywords: Knee brace; biomechanical footwear; exercise; RCT
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise therapy group (Active Comparator): (n = 40)
  Interventions: Other: Home-based exercise
- Knee brace and exercise group (Experimental): (n = 40)
  Interventions: Other: Home-based exercise; Device: Knee brace
- Footwear device group (Experimental): (n = 40)
  Interventions: Device: Biomechanical footwear device

INTERVENTIONS:
Other: Home-based exercise — Home-based exercises three times per week.
  Arms: Exercise therapy group; Knee brace and exercise group
Device: Knee brace — Progressive use of knee brace each day during activities of daily living.
  Arms: Knee brace and exercise group
Device: Biomechanical footwear device — Progressive use of footwear each day during activities of daily living.
  Arms: Footwear device group

SUMMARY:
This study investigates the effects of unloader knee brace, biomechanical footwear device and exercise therapy on pain, physical function and quality of life in patients with knee osteoarthritis. The aim is to find more effective treatment strategies to delay or prevent heavy knee replacement surgeries.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of exercising, and using a knee brace and exercising, and using of biomechanical footwear device on clinically important symptoms, physical function and quality of life in patients with osteoarthritis of the knee. The hypothesis is that the groups of using knee brace and biomechanical footwear can alleviate pain, improve physical function and quality of life more efficiently, than the group doing home exercises only.

The subjects (n = 120) will be randomized into three groups mentioned above, after which they will start to do exercises, or to use a knee brace and do exercises, or to use biomechanical footwear at home according to the instructions for 4 months. Physical function, symptoms and quality of life will be measured before and after 4-month intervention. In addition, at 12-month time point follow-up surveys will be addressed with regard to symptoms and quality of life, as well as to cost-effectiveness of the study.

ELIGIBILITY:
Inclusion Criteria:

* moderate or severe knee pain (>40mm on a VAS scale 0-100mm)
* radiographic knee osteoarthritis (Kellgren-Lawrence grades 1-3)
* age between 45 and 70 years

Exclusion Criteria:

* inflammatory joint disease
* acute (<6 months) knee trauma
* arthroscopic surgery in the past six months
* a planned knee replacement surgery or other planned surgical treatment of the knee
* knee injections in the past 3 months
* superficial wounds at the knee area
* arterial insufficiency
* severe varicosities
* impaired vision
* postural difficulties
* body-mass index (BMI) >35kg/m2
* fibromyalgia
* rheumatoid arthritis or other active rheumatoid inflammatory disease.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline Pain intensity at 4 months: VAS | 4 months
  Visual Analog Scale for Pain (score of 100 mm). No pain (score of 0), worst imaginable pain (score of 100).

SECONDARY OUTCOMES:
Change from baseline clinical symptoms at 4 months. | 4 months
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)-questionnaire evaluates the condition of patients with knee osteoarthritis including pain, stiffness and physical function. In the subscale of pain (score range 0 - 500), stiffness (score range 0 - 200), and functional limitation (score range 0 - 1700) lower values represent a better outcome. In order to normalize each score on 0 - 100 scales, the following correction factors are used: pain 0.20, stiffness 0.50, functional limitation 0.059.
Change from baseline Health-Related Quality of Life at 4 months: SF-36 | 4 months
  The SF-36-Item Health Survey measures Health-Related Quality of Life. The SF-36 is a multi-item scale assessing eight health concepts: 1) limitations in physical activities, 2) limitations in social activities, 3) limitations in usual role activities, 4) bodily pain, 5) general mental health, 6) limitations in usual role activities, 7) vitality, and 8) general health perceptions, with scores for each dimensions ranging from 0 (poor health) to 100 (good health).
Change from baseline isometric knee extension and flexion forces at 4 months. | 4 months
  Will be measured with dynamometer
Change from baseline walking speed gait parameter at 4 months. | 4 months
  Walking speed (cm/sec) will be measured by the instrumented walkway system (GAITRite mat).
Change from baseline cadence gait parameter at 4 months. | 4 months
  Cadence (steps per minute) will be measured by the instrumented walkway system (GAITRite mat).
Change from baseline stride length gait parameter at 4 months. | 4 months
  Stride length, i.e., the distance between 2 successive placement of the same foot (cm) will be measured by the instrumented walkway system (GAITRite mat).
Change from baseline step length gait parameter at 4 months. | 4 months
  Step length, i.e., the distance measured from the heel point of one foot to the heel point of the other foot (cm) will be measured by the instrumented walkway system (GAITRite mat).
Change from baseline stance time and % stance gait parameter at 4 months. | 4 months
  Stance time (sec) and % stance will be measured by the instrumented walkway system (GAITRite mat).
Change from baseline swing time and % swing gait parameter at 4 months. | 4 months
  Swing time (sec) and % swing will be measured by the instrumented walkway system (GAITRite mat).
Change from baseline 40 m Fast-paced Walk Test at 4 months. | 4 months
  A fast-paced walking test that is timed over 4 x 10m for a total 40 m
Change from baseline Stair Ascend/Descend Test at 4 months. | 4 months
  The time (sec) it takes to ascend and descend a flight of stairs. The total time to ascend and descend steps (negative number indicates better performance) will be recorded and reported
Change from baseline 30s Timed Chair Stand Test at 4 months. | 4 months
  The maximum number of chair stand repetitions possible in a 30 second period. The total number of chair stands (up and down equals one stand) completed in 30 seconds will be reported.
Change from baseline knee range of movement at 4 months. | 4 months
  Will be measured with goniometer
Change from baseline physical activity at 4 months. | 4 months
  The short form of International Physical Activity (IPAQ-SF) questionnaire measures data on Health-Related Physical Activity. The IPAQ-SF Records the activity of four intensity levels (vigorous-intensity, moderate-intensity, walking, sitting) for the last 7 days. Results are reported as a continuous variable (MET minutes a week). To calculate MET minutes a week the MET value given (walking = 3.3, moderate activity = 4, vigorous activity = 8) is multiplied by the minutes the activity was carried out and again by the number of days that the activity was undertaken. To get total MET minutes of physical activity a week, the MET minutes achieved in each category are added together. Higher MET-values represent better outcome.
Change from baseline cost-utility at 4 months. | 4 months
  Will be measured with the items of the SF-6D questionnaire, which in turn can be converted from the items of the SF-36 questionnaire. The SF-6D score varies from 0 to 1, 0 representing worst health cost-utility and 1 best health utility.

CONTACTS AND LOCATIONS:
Overall Officials: Jari Ylinen, Ph.D., M.D., Principal Investigator — Central Finland Hospital District; Arja Häkkinen, Ph.D., Study Chair — Central Finland Hospital District; Konsta Pamilo, M.D., Study Chair — Central Finland Hospital District; Ari Heinonen, Ph.D., Study Chair — University of Jyväskylä, Finland; Joost Dekker, Ph.D., Study Chair — VU University Medical Center, Amsterdam, Netherlands; Jari Arokoski, Ph.D, M.D., Study Chair — University of Eastern Finland
Locations (1):
- Central Finland Central Hospital, Jyväskylä, Finland

IPD SHARING:
Plan to Share IPD: No